CLINICAL TRIAL: NCT05049707
Title: Does Perioperative Intravenous Magnesium Affect Postoperative Quality of Recovery in Elective Craniotomy Surgery Patients?
Brief Title: Does Perioperative Intravenous Magnesium Affect Postoperative Quality of Recovery in Craniotomy Surgery Patients?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Kevin Min, Assistant Professor of Anesthesiology, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: #21D.124
Record Dates: First submitted 2021-08-31; First posted 2021-09-20 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Brain Tumor; Surgery
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The control arm will receive an equivalent volume of normal saline as the treatment group
  Interventions: Other: Placebo
- IV magnesium (Experimental): We will randomize patients in the treatment group to receive either a 50 mg/kg bolus of intravenous magnesium preoperatively followed by a magnesium infusion of 15mg/kg/hr, to be given after intraoperative neuromonitoring staff have been able to record baseline neurological data.
  Interventions: Drug: IV magnesium sulfate

INTERVENTIONS:
Drug: IV magnesium sulfate — 15 grams magnesium in 500 cc normal saline delivered at a rate of 15 mg/kg/hr
  Other Names: Magnesium Sulfate IV
  Arms: IV magnesium
Other: Placebo — 500 cc normal saline delivered in equivalent rates as the treatment group
  Arms: Control

SUMMARY:
Perioperative pain management for craniotomy patients may be challenging because the commonly used agents such as opioids, gabapentin, and dexmedetomidine also cause sedation, which can confound the neurological exam and can lead to respiratory depression and increased intracranial pressure. Preoperative intravenous magnesium boluses and infusions have previously been established as an effective, nonsedating analgesic that can reduce opioid consumption 25-30% up to 48 hours postoperatively.

However, intravenous magnesium has not seen widespread use in craniotomy patients due to concerns for interference with the neurological monitoring that commonly occurs in these cases. Intravenous magnesium given as a bolus preoperatively or as a constant infusion may avoid these problems and has never been investigated.

The goal of this study is to compare intravenous magnesium given preoperatively and intraoperatively to placebo in adult elective craniotomy patients to improve quality of recovery postoperatively, and evaluate safety and tolerability. Secondary endpoints will include evaluating for pain, sedation, agitation, blood pressure, and opioid consumption postoperatively.

DETAILED DESCRIPTION:
The study is a prospective, randomized, controlled, and double-blinded clinical trial comparing clinical outcomes of craniotomy patients who a magnesium infusion of 15mg/kg/hr to a placebo group of patients who will receive a saline bolus and infusion of equivalent volume starting at surgical closure and continuing for 15 hours. The sample size calculations are based on an effect size 24 point increase in Quality of Recovery-40 Questionnaire scores from a previous randomized control trial featuring the same bolus and infusion regimen as this trial. Investigators, patients, and providers will be blinded. Patients over the age of 18 undergoing elective craniotomy surgery will be enrolled.

The study population will consist of patients undergoing elective craniotomy surgery. The inclusion criteria consists of patient age 18-85, ASA (American Society of Anesthesiologists) Physical Status Classification 1-3, with Glasgow Coma Scale (GCS) of 15 with adequate english comprehension. Exclusion criteria includes pregnant or nursing patients, patients with known allergies to any of the study drugs, patient's refusal, patients with a history of cirrhosis, chronic kidney disease stage 3 or higher, known history of substance abuse, neuromuscular disease or heart block.

ELIGIBILITY:
Inclusion Criteria:

* patient age 18-85
* ASA (American Society of Anesthesiologists) Physical Status Classification 1-3
* Glasgow Coma Scale (GCS) of 15
* Adequate english comprehension

Exclusion Criteria:

* pregnant or nursing patients
* patients with known allergies to any of the study drugs
* patient's refusal
* patients with a history of cirrhosis
* chronic kidney disease stage 3 or higher
* known history of substance abuse
* history of neuromuscular disease
* history of heart block

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery Questionnaire 40 | Postoperative days 0-2
  Validated measure of postoperative quality of recovery

SECONDARY OUTCOMES:
Hypertension Postoperative | postoperative days 0-2
  systolic blood pressure > 160
Postoperative Hyperglycemia | Postoperative days 0-2
  glucose > 180
Complications Possibly Related to Intraoperative Neuromonitoring | postoperative days 0-2
  We will monitor for rates of complications postoperatively, noting whether or not they could have been detected by intraoperative neuromonitoring
Shivering | First 2 hours in the postoperative care unit or intensive care unit
  Bedside Shivering Scale

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Min, MD, Principal Investigator — Thomas Jefferson University

IPD SHARING:
Plan to Share IPD: No